CLINICAL TRIAL: NCT03224858
Title: Does a Clinic Based Complex Care Coordination Intervention Improve Patient Quality Outcomes in an Underserved Clinic Population? The Streamlined, Unified, Meaningfully Managed Interdisciplinary Team (SUMMIT) Ambulatory ICU Study
Brief Title: Ambulatory ICU Study for Medically and Socially Complex Patients
Acronym: SUMMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Brian L Chan, assistant professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 15285
Record Dates: First submitted 2017-06-28; First posted 2017-07-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Health Services; Comorbidity; Primary Health Care
Keywords: Patient-Centered Care; Comorbidity

STUDY DESIGN:
Intervention Model Description: This is a pragmatic "wait-list" control design. Participants will be consented and baseline survey administered after which patient will be randomized by computer generated algorithm into 2 arms: immediate or 6-month 'wait-list.' Immediate group will start intervention and be followed at 6 month intervals for 12 months. 'Wait-list' group will resume usual care for 6-months, after which they will cross-over to the intervention group for 12 months.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, care providers, investigator, and initial trained research assistant will be blinded initially during consent and baseline interview survey procedures. Once, randomization has occurred, the participants, care provider, investigator, and subsequent outcomes assessor will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SUMMIT intervention group (Experimental): This group will transfer primary care to the SUMMIT team, which consists of: 1 primary care provider, 1 clinical nurse, 1 team manager, 2 care-coordinators, 2 behavioralists, 1 clinical pharmacist. This interdisciplinary team will have reduced patient panel load and increased flexibility in time and scheduling in order to foster trust and continuity with the patient with a goal of decreasing treatment burden and increasing patient capacity. Specific activities that participants will receive include: 1) comprehensive initial intake and care plan development that incorporates patient goal setting; 2) flexible scheduling of appointments with outreach; 3) transitional care coordination; 4) built-in behavioural counselling and case management; 5) regular review of care plan by team members.
  Interventions: Other: SUMMIT intervention
- enhanced usual care group (Active Comparator): This group will continue to receive primary care as usual for 6 months. This includes care provided by the patient's existing primary care provider, access to a clinic's Health Resilience outreach worker, mental health consultation, and other services provided by usual care. After 6 months, the baseline survey is administered and the participant will transfer care to the intervention as described above in the SUMMIT intervention group.
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Other: SUMMIT intervention — See description in experimental arm.
  Other Names: intensive primary care team, complex care team
  Arms: SUMMIT intervention group
Other: Enhanced usual care — See description in active comparator arm.
  Other Names: usual care
  Arms: enhanced usual care group

SUMMARY:
This is a prospective randomized wait-list control study to determine whether a stand-alone, co-located team of physician, mental health behaviorist, and care coordinators with decreased panel size (aka "intensive primary care") will reduce inpatient and emergency care utilization, inpatient costs of care, and improve patient activation and experience for medically and socially complex patients, compared to enhanced usual care at 6 and 12 months. Participants with multiple co-morbidities, and meet utilization criteria will have the opportunity to enroll; half the participants will start the intervention immediately, while half will continue enhanced usual care for 6 months before beginning the intervention.

DETAILED DESCRIPTION:
The goal of this study is to conduct an evaluation of an "Ambulatory-ICU" model of primary care for "high utilizer" patients with medical, behavioral, and social complexity. A small proportion of patients use > 50 % of healthcare resources. It is currently unknown what interventions can help reduce inappropriate utilization due to lack of studies with rigorous study design, particularly in patients with high rates of homelessness, mental illness and substance use. The use of high-risk teams for select patients is a promising model of primary care that removes barriers to accessing usual care services by centralizing medical and behavioral clinical services, promotes ability to outreach beyond the clinic, and promote continuity of care and trust-building between patient and provider teams.

This study will test the hypothesis that a stand-alone clinic based intervention of a multidisciplinary, co-located physician, mental health behaviorist, nursing, pharmacist, and care coordinators with reduced panel size, and focus on patient capacity building and decreasing treatment burden will improve health outcomes at 6 and 12 months in a low-income high utilizer population with history of homelessness.

Enhanced usual care comprises of care delivered at Old Town Clinic (OTC) a Federally Qualified Health Center (FQHC) that is modeled on the Patient Centered Medical Home (PCMH) model. Patients have a designated primary care physician and care team with access to chronic disease education, mental health, social work, and substance abuse programs through referral system. In addition, participants thought to have difficulty engaging in primary care have access to a Health Resilience Specialist, a community health worker intervention who conducts outreach and assists the patient in care navigation.

ELIGIBILITY:
Inclusion Criteria:

• One or more of the following medical diagnoses:

* congestive heart failure
* uncontrolled diabetes
* end stage liver disease
* chronic kidney disease (stage III or higher)
* chronic obstructive pulmonary disease (group C or D)
* chronic or severe soft tissue infections or ulcers
* osteomyelitis
* failure to thrive

And/OR:

• One or more of the following behavioral health diagnoses:

* psychotic disorder
* mood disorder
* post-traumatic stress disorder
* active substance use disorder

And/OR

• One or more of the following utilization patterns:

* 1+ medical hospital admission in prior 6 months
* frequent missed appointments (cancel or no-show for >5 primary care or specialty appointments in previous 12 months

Exclusion Criteria:

* Non-English speaking
* Patients on hospice, nursing home, rehabilitation, or other institutional or long term care facility
* Inability to consent (as demonstrated by teach back of the consent process)
* Diagnosis of metastatic brain cancer
* Inability to participate in follow up phone due to aphasia, severe hearing impairment, or lack of access to telephone

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-09-27 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Medical Hospitalizations | 6 months
  Administrative data will be used to determine hospital admissions
Emergency Care visits | 6 months
  Administrative data will be used to determine Emergency Department (ED) visits over study period
Primary care utilization | 6 months
  Clinic administrative data will be used to determine primary care visits over study period
Patient Activation Measure (PAM) | 6 months
  Study survey of the PAM measure is a validated instrument to assess patient self-efficacy
Patient Experience (ambulatory CAHPS) | 6 months
  Study survey of patient reported assessment of patient experience

SECONDARY OUTCOMES:
Life Chaos | 6 months
  Study survey of a validated instrument to assess self-reported life chaos
inpatient costs of care | 6 months
  claims data for patients will be used to determine costs of inpatient care
inpatient average length of stay | 6 months
  Administrative data will be used to determine average length of stay each hospitalization
Functional status using Short Form (SF)-12 survey | 6 months
  patient reported survey of functional status
number of falls | 6 months
  Study survey with question asking how many falls over the last 6 months
Edmonton Symptom Assessment Scale (ESAS) palliative measure | 6 months
  Study survey with one question from the ESAS questionaire
Medical Hospitalizations | 12 months
  Administrative data will be used to determine hospital admissions
Emergency Care visits | 12 months
  Administrative data will be used to determine ED visits
Patient Activation Measure (PAM) | 12 months
  Study survey of the PAM measure is a validated instrument to assess patient self-efficacy
Primary care utilization | 12 months
  Clinic administrative data will be used to determine primary care visits over study period

CONTACTS AND LOCATIONS:
Overall Officials: Brian Chan, MD, Principal Investigator — Assistant Professor
Locations (1):
- Central City Concern, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
upon request, the investigators can share de-identified, cleaned IPD for other researchers.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Chan B, Edwards ST, Devoe M, Gil R, Mitchell M, Englander H, Nicolaidis C, Kansagara D, Saha S, Korthuis PT. The SUMMIT ambulatory-ICU primary care model for medically and socially complex patients in an urban federally qualified health center: study design and rationale. Addict Sci Clin Pract. 2018 Dec 14;13(1):27. doi: 10.1186/s13722-018-0128-y. PMID 30547847
- [Background] Chan B, Hulen E, Edwards S, Mitchell M, Nicolaidis C, Saha S. "It's Like Riding Out the Chaos": Caring for Socially Complex Patients in an Ambulatory Intensive Care Unit (A-ICU). Ann Fam Med. 2019 Nov;17(6):495-501. doi: 10.1370/afm.2464. PMID 31712287
- [Derived] Chan B, Cook R, Levander X, Wiest K, Hoffman K, Pertl K, Petluri R, McCarty D, Korthuis PT, Martin SA. Buprenorphine discontinuation in telehealth-only treatment for opioid use disorder: A longitudinal cohort analysis. J Subst Use Addict Treat. 2024 Dec;167:209511. doi: 10.1016/j.josat.2024.209511. Epub 2024 Sep 5. PMID 39243979
- [Derived] Chan B, Edwards ST, Srikanth P, Mitchell M, Devoe M, Nicolaidis C, Kansagara D, Korthuis PT, Solotaroff R, Saha S. Ambulatory Intensive Care for Medically Complex Patients at a Health Care Clinic for Individuals Experiencing Homelessness: The SUMMIT Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2342012. doi: 10.1001/jamanetworkopen.2023.42012. PMID 37948081